CLINICAL TRIAL: NCT05873894
Title: Acute Pain Oscillation in Electroencephalographic Monitoring Under General Anaesthesia: Characterisation of EEG Patterns Secondary to Pain
Brief Title: Acute Pain Oscillation in Electroencephalographic Monitoring Under General Anaesthesia
Acronym: EEGpain
Status: Recruiting | Type: Observational
Sponsor: Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Carolina Soledad Romero Garcia, MD, PhD, Professor, Hospital General Universitario de Valencia
Other Study IDs: 31/2020
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EEG — EEG recordings and analysis. Sensory evoked potentials analysis Motor evoked potentials studies

SUMMARY:
Chronic pain is an undesirable condition that impacts predominantly quality of life at all levels. Chronic pain might occur in healthy young patients when acute postoperative pain is undertreated and persists in time. There are some indexes in the market to evaluate pain, but they assess mainly parasympathetic activity. Hence, it´s a measure of the physiological response to pain, which is still a not well-defined concept. Patients under General Anesthesia might be experimenting unnoticed pain as there is no direct standard method to measure it in clinical practice. This study aims to detect brain oscillatory activity in the intraoperative setting in four situations; awake-no pain, awake-pain, sleep-no pain, and sleep-pain. Pain can be assessed by studying the local and global dynamics of brain activity. A promising upcoming measure of pain could be implemented in clinical practice to detect and treat pain.

DETAILED DESCRIPTION:
This is a pilot study of the presence of neural oscillations during acute pain while awake and in the anesthetized patient with neurophysiological monitoring during a neurosurgery surgical intervention analyzed by electroencephalography.

After the patient's consent, the electroencephalogram is placed in the awake patient and a small painful stimulus is performed based on the channeling of a second venous access. In turn, a recording of the EEG waves is made in order to identify similar neuronal waves during the surgical procedure once the patient is under general anesthesia.

The reason for this intervention is to have a baseline record of each patient without interfering with the oscillations of the different drugs used during total intravenous anesthesia used in these procedures. Normally, after general anesthesia, between 3 and 6 electrodes would be placed on the scalp and 10 electrodes would be placed to carry out this work.

After the intervention, a telephone survey will be carried out on postoperative pain at 3 months and a year.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients that undergo schedule neurosurgery with neurophysiological monitorisation.
* American Society of Anaesthesiologist physical status (ASA) I-IV.

Exclusion Criteria:

* Pregnancy
* Obstructive hydrocephaly with or with a derivative catheter.
* Patients with neurostimulator
* Emergency surgery.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with anaesthesia and eeg monitoring
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Oscillations related to pain in the EEG | since start of surgery until the end
  The main objective is the characterization and evaluation of the neural oscillations in the EEG that occur in the anesthetized patient when acute intraoperative pain occurs during monitoring by neurophysiology in neurosurgery.
  The current procedure includes patient monitoring with neurophysiology electrodes at muscle level and EEG for proper mapping of the functions to be explored when the patient is under the effects of general anesthesia.
  To carry out this work, it would be necessary to monitor the EEG with the patient awake, since it is intended to look for the characteristic neural oscillations at the moment in which the second peripheral venous line is cannulated.

SECONDARY OUTCOMES:
Incidence of Chronic pain | after surgery until 1 year post surgery
  1. Develop an objective scale of pain in the patient under general anesthesia.
  2. Evaluate the degree of pain 3 months after surgery using the visual analogue scale in the operated patients or/and Pain Detect Questionnarie .
opiod consumption | during surgery until 1 year post surgery
  During the intraoperative phase we will base ourselves on the equivalence between the use of intravenous fentanyl or oxycodone and intravenous morphine. For the subsequent evaluation of opioid consumption one year after surgery, we will base ourselves on the conversion tables to oral morphine.

CONTACTS AND LOCATIONS:
Locations (1):
- CHGUV, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Research board decision was not to share Individual Participant Data